CLINICAL TRIAL: NCT03771716
Title: Rhythm Experience and Africana Culture Trial II
Brief Title: Rhythm Experience and Africana Culture Trial
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kirk Erickson, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY19020263; 1R01AG060741-01 (NIH)
Record Dates: First submitted 2018-11-30; First posted 2018-12-11 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Performance; Brain Structure

STUDY DESIGN:
Intervention Model Description: 180 African American older adults between the ages of 60-80 will be randomly assigned to one of two groups: African Dance or Africana Culture. Both groups will meet 3 times per week for 1 hour over a period of 6-months. Cognitive and brain metrics will be assessed at baseline and following the completion of the intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Neither the investigator, nor outcomes assessors will know participants' group assignments. Participants will be instructed to refrain from speaking about their group's activities when visiting the lab for follow-up assessment. In addition, special care was taken to ensure that non-blinded laboratory staff (e.g., staff member notifying participants of their group assignments, staff monitoring the intervention classes) are not located in the same proximity in the laboratory, further preventing accidental unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- African Dance (Experimental): This is the experimental group. Dance classes will be held 3 times per week for 1 hour. Participants will learn traditional Africana dance moves and sequences.
  Interventions: Behavioral: African Dance
- African Cultural Immersion (Active Comparator): This is the active control group. Participants will participate in a variety of educational activities related to African Culture, including traditional cooking, lectures, crafts, music and films. They will meet 3 times per week for the same duration as the Dance group. However, they will not participate in aerobic activity during the classes, and most activities will be conducted in a seated position.
  Interventions: Behavioral: African Cultural Immersion

INTERVENTIONS:
Behavioral: African Dance — Basic principles and guidelines for exercise programming will be followed including adequate warm-up and cool-down, progressive and gradual increments in duration, and instruction regarding avoidance of physical activity (PA) related injury. The African dance group will receive moderate intensity dance 1 hour per day, twice per week, for 6 months. The prescribed intensity will begin at light to moderate and progress to a moderate to high intensity level. Frequent assessment of heart rate and ratings of perceived exertion will ensure appropriate levels of intensity during each dance session. Levels of exertion during the dance will be prescribed and monitored based on baseline assessments of heart rate and cardiorespiratory fitness.
  Other Names: Dance Group
  Arms: African Dance
Behavioral: African Cultural Immersion — The Culture group will participate in activities, including cooking, art and games, music, traditional crafts, and lectures and discussions about other aspects of Africana culture and customs. Topics will vary from session to session to maintain interest and engagement. The sessions will be held in a small group format and will be lead my personnel with training in each topic. Participants will meet 1 hour per day, 3 times per week, for 6 months.
  Other Names: Culture Group
  Arms: African Cultural Immersion

SUMMARY:
REACT is a randomized intervention to examine the benefits of African Dance as a method to increase physical activity behaviors in older adults. In this 6- month intervention, older African Americans will be randomly assigned to either an African Dance or an Africana Culture class. Both before and at the completion of the intervention, the investigators will collect a comprehensive neuropsychological battery and MRI scans of brain health and function to better study how physical activity influences neurocognitive health in African Americans.

DETAILED DESCRIPTION:
Aim 1: Examine whether the African Dance intervention improves cognitive performance compared to an educational control group. H1: The dance group will show cognitive improvements in a domain-specific fashion such that executive and memory functions will be enhanced more than other cognitive domains; Aim 2. Examine whether African Dance influences brain morphology, task-evoked neural responses, cerebral blood flow, and resting state connectivity. H1: It is predicted that African Dance will increase volume, white matter integrity, perfusion, and functional activation/connectivity in a regionally-specific fashion such that prefrontal and hippocampal areas will be more sensitive to the intervention than other brain regions. Aim 3. Explore potential physiological and socio-emotional mechanisms of the dance intervention. The investigators will collect measures of physical and psychosocial health such as waist circumference, blood pressure, blood glucose and lipid levels, mood, anxiety, depression, and loneliness and examine whether intervention-related changes to these measures mediate improvements in cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* self identifies race as African American
* between 60 and 80 years of age
* ambulatory without pain or the assistance of walking devices
* no history of falls or balance problems
* able to speak and read English
* available during the times classes are offered and able to make at least 80% of classes (e.g., no long-term travel plans)
* reliable means of transportation
* scores above the range on the Brief Telephone Interview for Cognitive Status (TICS) indicative of moderate to severe cognitive impairment (scores 21 or above)
* no diagnosis of a neurological disease or psychiatric conditions
* eligible to undergo MRI (not claustrophobic and no metal or history of injury involving metal).
* Fully vaccinated for coronavirus disease (COVID-19).

Exclusion Criteria:

* self identifies race as other than African American
* not between 60 and 80 years of age
* not ambulatory without pain or the assistance of walking devices
* history of falls or balance problems
* unable to speak and read English
* unavailable during the times classes are offered or unable to make at least 80% of classes (e.g., indicates long-term travel plans during intervention period)
* no reliable means of transportation
* scores in range on the TICS indicative of moderate to severe cognitive impairment (scores 21 or below)
* has a diagnosis of a neurological disease or psychiatric condition
* ineligible to undergo MRI (claustrophobic and/or metal in body or history of injury involving metal).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk I Erickson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | African Dance | African Cultural Immersion
Started | 75 | 76
Completed | 59 | 62
Not Completed | 16 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African Dance | African Cultural Immersion | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.23 (4.94) | 67.11 (4.58) | 67.17 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 127
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 71 | 74 | 145
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 74 | 71 | 145
  White | 0 | 0 | 0
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Cardiorespiratory fitness (VO2peak) [Mean (Standard Deviation); unit: mL/kg/min] | 16.45 (4.12) | 15.89 (3.83) | 16.17 (3.98)

OUTCOME MEASURES:

1. Primary Outcome: Flanker Performance
Description: A Flanker Inhibitory Control and Attention task will be administered at baseline, and then following the intervention (6 months). The main outcome from this task is the computed score from the NIH Toolbox, which reflects the participant's ability to inhibit responses to irrelevant information while focusing attention on a target stimulus. In each trial, participants make a directional response to a center arrow when the flanking arrows are arranged in congruent vs. incongruent direction from the center stimulus. The computed score combines accuracy and reaction time into a single performance metric, ranging from 0 to 10, with higher values indicating better performance. Group differences will be tested on this outcome.
Time Frame: Changes from baseline to 6-months
Population: All participants data were included, as we conducted intention-to-treat (ITT) analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | African Dance | African Cultural Immersion
Number analyzed (Participants) | 75 | 76
score on a scale | -0.1055 [-0.253 to 0.0421] | -0.0586 [-0.203 to 0.0857]

2. Secondary Outcome: Hippocampal Volume (mm3)
Description: Structural scans will be collected at baseline as well as following the intervention. Hippocampal volume will be calculated in mm3. The investigators will examine group differences in size of the hippocampus following the intervention.
Time Frame: Changes from baseline to 6-months
Population: All participants data were included, as we conducted intention-to-treat (ITT) analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: cubic millimeters (mm³)
Arm/Group | African Dance | African Cultural Immersion
Number analyzed (Participants) | 75 | 76
cubic millimeters (mm³) | -7.57 [-107.28 to 92.14] | -59.71 [-149.78 to 30.36]

3. Other Pre Specified Outcome: Change in Cognitive Function
Description: Investigators are assessing change in cognitive function from baseline to 12 months. A comprehensive neuropsychological battery will be used that assesses 5 domains of cognitive function (Working Memory, Processing Speed, Episodic Memory, Attentional Control, and Visuospatial Function). We will perform a confirmatory factor analysis on the cognitive data and determine whether the exercise intervention influences performance as measured by these factors. There is no min and max values. These are generated from a confirmatory factor analysis that normalizes the scores around 0 (being the mean). As such, positive values reflect better performance and negative values reflect poorer cognitive performance. Since the scores are standardized we can calculate the changes in standard deviations - e.g., a shift of 0.5 would be an improvement of ½ standard deviation in performance based on the sample average.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Medication Use
Description: We will be recording all prescribed and over-the-counter (OTC) medications that the study participant is currently taking and will examine whether the intervention effects vary as a function of medication use.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Cardiorespiratory Fitness
Description: The investigators will conduct a sub-maximal fitness test before and after the intervention in order to calculate each participant's fitness level (via estimated VO2 max). The investigators will examine group differences in fitness following the intervention.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Functional Fitness
Description: Senior Fitness Test will be used to measure various aspects of fitness - e.g., balance, flexibility, strength. We will examine whether the exercise intervention improves any marker of fitness.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Actigraphy Steps Per Day
Description: The investigators will collect objective physical activity levels via wrist-worn accelerometers every 6 weeks throughout the intervention. Steps per day will be a primary outcome from the actigraphy. The investigators will examine changes in physical activity over the intervention.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Exercise Frequency
Description: Exercise frequency will be measured using Actigraph Link physical activity monitoring device. This device is small and lightweight. It is worn around the non-dominant wrist(touching the skin) for approximately 7 days during all waking and sleeping hours. We will examine whether the intervention altered this measure of daily activity.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Exercise Intensity
Description: Exercise intensity will be measured using the Actigraph Link physical activity monitoring device. This device is small and lightweight. It is worn around the non-dominant wrist (touching the skin) for approximately 7 days during all waking and sleeping hours. We will examine whether the exercise intervention altered amount of time spent in moderate-to-vigorous activities during daily life.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Exercise Duration
Description: Exercise duration will be measured using Actigraph Link physical activity monitoring device. This device is small and lightweight. It is worn around the non-dominant wrist (touching the skin) for approximately 7 days during all waking and sleeping hours.. The duration is measured in minutes. We will examine whether the exercise intervention altered amount of time spent in moderate-to-vigorous activities during daily life.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Weight
Description: Participants will be weighed on a calibrated stadiometer both before and after the intervention. The investigators will examine percent changes in body weight in the groups before and after the intervention.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Hippocampal Subfield Volumes
Description: MRI will be used to measure volumetric changes in hippocampal subfields.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in White Matter Lesions
Description: MRI will be used to measure changes in white matter microstructure in relation to the intervention.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in White Matter Diffusion Properties
Description: MRI will be used to measure changes in white matter microstructure in relation to the intervention.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Cerebral Blood Flow
Description: MRI will be used to measure changes in cerebral blood flow. Total cerebral blood flow changes over the course of the intervention will be evaluated.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Resting State Brain Activity
Description: MRI will be used to measure changes in resting state brain function. We will examine whether the intervention alters resting state connectivity metrics.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Task-evoked Relational Memory Brain Activity
Description: MRI will be used to measure changes in encoding and retrieval during a relational memory task.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Task-evoked Working Memory Brain Activity
Description: MRI will be used to measure changes in brain activity task-evoked patterns using an N-back working memory task.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Cortical Thickness
Description: MRI will be used to measure average cortical thickness over the course of the intervention.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Changes in Blood Levels of Cholesterol
Description: The investigators are collecting data on changes in blood biomarkers including levels of cholesterol, low-density lipoprotein (LDL), very low-density lipoprotein (VLDL), high-density lipoprotein (HDL), and triglycerides.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Blood Levels of Glucose
Description: The investigators will examine whether changes in markers of insulin resistance change over the course of the intervention and whether these changes mediate neurocognitive outcomes.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Change in Blood Levels of Hemoglobin
Description: The investigators are collecting data on changes in average blood sugar levels (HbA1C)
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Socioeconomic Status (SES) Composite
Description: Combining information from the MacArthur questionnaire to develop Social Economic Status of participants, we will examine whether the effectiveness of the intervention varied by SES levels of the participants. The SES composite is generated using a confirmatory factor analysis of various SES indicators - e.g., income, debt, savings, etc. The scores are normalized so that 0 is the average for the sample, higher numbers reflect higher SES, and lower numbers indicate lower SES.
Time Frame: Baseline
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Health History & Lifestyle Habits
Description: Health History assesses medical history and lifestyle habits such as alcohol and tobacco use. We will examine whether any neurocognitive outcomes vary as a function of these health conditions and behaviors.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Depression
Description: The investigators are collecting a questionnaire measuring depressive symptoms, the Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D is a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. The questionnaire will be administered at baseline as well as at the 6-month followup.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Loneliness
Description: The investigators are collecting a questionnaire measuring self-perceived loneliness, the University of California Loneliness Scale (UCLALS). This is a 20-item scale in which participants rate frequency of feelings of loneliness and social isolation on a 4 point scale ranging from "never" to "often". A total score is computed which can range from 20- 80. Higher scores indicate more loneliness. The questionnaire will be assessed at baseline as well as at the 6-month followup.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Mindfulness
Description: The Mindful Attention Awareness Scale (MAAS) assesses a core characteristic of mindfulness mainly open or receptive awareness of and attention to what is taking place in the present. We will examine whether the exercise intervention altered measures of mindfulness. Score scale runs 15-90 with higher scores reflecting more mindfulness.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Positive and Negative Affect
Description: The Positive and Negative Affect Schedule (PANAS) is used to measure mood and emotion. It is comprised of 20 items, with 10 items measuring positive affect (e.g., excited, inspired) and 10 items measuring negative affect (e.g., upset, afraid). Each item is rated on a five-point Likert scale. Positive affect scores range from 10 to 50, and negative affect scores range from 10 to 50.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

29. Other Pre Specified Outcome: State Trait Anxiety Inventory (STAI)
Description: The STAI is a validated 20 item self-report assessment which includes separate measures of state and trait anxiety. The inventory includes 40 items on a 4-point Likert scale. Higher scores indicate higher levels of anxiety.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Perceived Pain
Description: The McGill Pain Questionnaire is used to evaluate a person's perception of pain. It can be used to monitor the pain over time and to determine the effectiveness of any intervention. We will examine whether the intervention alters perceptions of pain in late adulthood. Score scale runs 0-45 with higher values meaning more pain.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Perceived Fatigability
Description: The Pittsburgh Fatigability Scale assesses self-report whole-body physical and mental tiredness related to activities of fixed intensity and duration in adults age ≥60. The scale includes 10 items, each measured on a 5-point Likert scale for a total score of 0-50. Higher scores indicate higher fatigability.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Levels of Inactivity
Description: Sitting Time Questionnaire scores how much time is spent sitting during 5 different events on a weekday and weekend day. We will examine whether participating in the intervention alters amount of time spent sitting. Calculate weekly minutes with higher values in minutes = more sedentary (sitting time)
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Lifestyle Physical Activities
Description: The Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire assesses self-report weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults. It includes activities of various intensities (from light to vigorous) such as walking, running, hiking, swimming, bicycling, dancing, tennis, aerobics, yoga/tai chi, gardening, and housework. For each activity, the following measures are scored: frequency per week, hours per week, estimated caloric expenditure per week, and mets/kg/week.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Perceived Sleep Quality
Description: Pittsburgh Sleep Quality Index (PSQI) will be used to assess perceived sleep quality. We will examine whether the exercise intervention alters perceived sleep quality. All components have score range 0-3 with lower number equal to better sleep quality.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Exercise Self-Efficacy
Description: The investigators will use the Exercise Self-Efficacy Scale (EXSE) to assess belief in the ability to continue exercising three times a week at a moderate intensity for 40 plus minutes a session into the future. We will examine whether this measure predicts long-term adherence outcomes. Score scale runs 0-100 with higher values = higher confidence to continue to exercise (3X's week for 40 + minutes) in the future 8 weeks
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Barriers to Exercise (BARSE)
Description: BARSE questionnaire assess degrees of confidence that one could exercise despite a variety of limitations such as during bad weather, while on vacation, etc. This scale was designed to tap subjects' perceived capabilities to exercise three times per week for 40 minutes over the next two months in the face of commonly identified barriers to participation. We will examine whether measures of barriers predicts adherence and compliance to the intervention. Scale 1-100, higher values = higher level of perceived capability to overcome barriers to exercise
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Social Provisions
Description: Social Provisions Scale (SPS):A 24-item scale assessing six relational provisions: attachment, or emotional support; social integration, or network support; reassurance of worth, or esteem support; reliable alliance, or tangible aid; guidance, or informational support; and the opportunity of nurturance.The items were modified for the exercise setting. For example, one of the statements used to assess social integration was "I feel part of the exercise group". We will examine whether social provisions relates to adherence to the intervention. Each subscale has range of 4 - 16 with total score range 24 - 96, higher values = higher social relationship (ppt. is receiving that provision)
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Physical Activity Self-Regulation
Description: Physical Activity Self-Regulation Scale, 12-item version (PASR-12): (PASR-12 FORM) A 12-item version of a popular 43-item self-regulation scale. Participants were asked to rate how often they used each strategy on a scale from 1 (never) to 5 (very often). We will examine whether measures of self-regulation predicts adherence and compliance to the intervention. Each subscale has range of 2 - 10, higher scores = greater use of self-regulation strategies. Summary score has range of 12 - 60
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Perceived Weight Discrimination
Description: Hunger and Major (2015) developed a perceived weight discrimination scale based on a widely-used measure of racial discrimination. Participants respond to five items (e.g., "In the past 12 months, how often other people treated you unfairly because of your weight?") on 0 (never) to 4 (all the time) scales. We will examine whether the exercise intervention modified measures of perceived weight discrimination.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Perceived Health & Quality of Life
Description: The Short Form Health Survey (SF-36) taps into eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. We will examine whether the exercise intervention modified measures of health related quality of life. Each concept has a score range of 0-100 with higher scores equal to more favorable health traits.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Life Satisfaction
Description: We will use the Satisfaction with Life Scale (SWLS) as a global cognitive judgement of study participants life satisfaction. We will examine whether the exercise intervention altered SWLS measures. Total score range is 5 -35 with higher scores equal to greater satisfaction with life.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Subjective Cognitive Performance
Description: Everyday Cognition (ECOG)(Short version) measures subjective cognitive performance. We will examine whether the intervention alters this subjective/perceived level of cognitive function. Score range is 1 - 4 with lower scores equal to better daily function.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Perceived Cognitive Abilities
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Applied Cognition: (Abilities) This is a brief self-report of perceived cognitive abilities for daily functioning. We will examine whether the intervention alters this subjective/perceived level of cognitive function. Scale 8-40, assess ppt. perceived functional abilities in regard to cognitive tasks. Higher value = higher self-perceived ability in cognition.
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Perceived Cognition for Daily Life
Description: PROMIS Applied Cognition: (General Concerns) This is a brief self-report of perceived difficulties with cognition for daily functioning. We will examine whether the intervention alters this subjective/perceived level of cognitive function. Scale 8-40. Lower score = less cognitive concerns
Time Frame: Changes from baseline to 6-months
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Black Identity
Description: The Multidimensional Model of Racial Identity (MMRI) is a model that identifies four dimensions of African American racial identity: salience, centrality, regard, and ideology. We will examine whether racial identity acts as mediator to cognitive performance post-intervention.
Time Frame: 6-month post
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Race-Related Stress
Description: The Index of Race-Related Stress (IRRS) is one of the most commonly used measures to assess race-related stress among Black Americans. We will examine whether racial identity acts as mediator to cognitive performance post-intervention.
Time Frame: 6-month post
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | African Dance | African Cultural Immersion
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 4/75 | 5/76
Other Adverse Events (participants affected / at risk) | 12/75 | 10/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | African Dance (N=75) | African Cultural Immersion (N=76)
Nephrolithiasis (Surgical and medical procedures) | 1 | 2
Hip replacement (Surgical and medical procedures) | 0 | 2
Fall; Multiple traumatic injuries (Injury, poisoning and procedural complications) | 3 | 0
Eye Surgery (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | African Dance (N=75) | African Cultural Immersion (N=76)
abnormal blood pressure (Vascular disorders) | 3 | 4
Ankle/Muscle injury (Musculoskeletal and connective tissue disorders) | 2 | 3
Gastro-Intestinal (Gastrointestinal disorders) | 2 | 0
Incidental finding (General disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Allergy reaction (Immune system disorders) | 0 | 1
Skin disorder (Vascular disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT03771716/Prot_SAP_000.pdf